CLINICAL TRIAL: NCT00491452
Title: Repair of Ischemic Mitral Regurgitation: Comparison Between Flexible and Rigid Annuloplasty Rings
Acronym: IMR2
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: ISCH-MR1
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Mitral Regurgitation
Keywords: Ischemic MR; Annuloplasty
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Mitral valve repair for ischemic mitral regurgitation is performed primarily by annuloplasty. There is some degree of late failure, which may be due in part to the type of ring employed. We want to compare late results with mitral valve annuloplasty using flexible vs rigid annuloplasty rings.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing CABG with Mitral valve repair for ischemic MR

Exclusion Criteria:

* Other valve procedures

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing CABG with Mitral valve repair for ischemic MR
Sampling Method: Non-Probability Sample
Dates: Start 2007-04; Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuli Silberman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel